CLINICAL TRIAL: NCT06771180
Title: Daratumumab, Bortezomib, Cyclophosphamide, and Dexamethasone Therapy for Patients with Rare Monoclonal Gammopathies of Renal Significance
Brief Title: Dara-BCD for Rare MGRS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Dr, Peking University People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB134-002
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Monoclonal Gammopathy of Renal Significance (MGRS)
Keywords: PGNMIDs; LCPT; TMA; CGGN; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dara-CyBorD (Experimental): Daratumumab Cyclophosphamide Bortezomib Dexamethasone
  Interventions: Drug: Dara-CyBorD

INTERVENTIONS:
Drug: Dara-CyBorD — Dara-CyBorD will be used for newly diagnosed PGNMID, OR LCPT, OR TMA OR CGGN.

SUMMARY:
This is an open-label, multicenter, phase 2 study in subjects with newly diagnosed proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMIDs), OR light chain proximal tubulopathy (LCPT), OR thrombotic Microangiopathy (TMA), OR cryoglobulinemic glomerulonephritis, (CGGN), treated with daratumumab, bortezomib, cyclophosphamide, and dexamethasone.

DETAILED DESCRIPTION:
The current study aims to investigate daratumumab, bortezomib, cyclophosphamide, and dexamethasone regimen in patients with newly diagnosed PGNMIDs, LCPT, TMA, CGGN. Approximately 10 subjects will receive primary therapy with daratumumab-CyBorD. The primary endpoint is overall complete hematologic response (CHR) rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PGNMIDs, OR LCPT, OR TMA, OR CGGN.
2. Evidence of clonal plasma cell in bone marrow.
3. ECOG 0,1,2
4. Neu≥ 1.0*10^9/L, HGB ≥70g/L, PLT ≥ 50*10^9/L.
5. Total bilirubin (TBil) ≤3×upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN;
6. Informed consent explained to, understood by and signed by the patient.

Exclusion Criteria:

1. Prior therapy for MGRS, with the exception of equal or less than 160 mg dexamethasone (or equivalent corticosteroid)
2. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma.
3. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
4. Severe or persistent infection that cannot be effectively controlled;
5. Presence of severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]); Patients with HIV infection or syphilis infection;
7. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Hematologic Complete Response at the completion of 6 cycles | 6 months
  Hematologic complete response requires absence of monoclonal protein by immunofixation electrophoreses of both serum and urine as well as a normal FLC ratio (FLCr). CR is considered when FLCr was altered in favour of the non-amyloidogenic, uninvolved FLC (uFLC), even though the ratio may not have been normalised.

SECONDARY OUTCOMES:
Rate of Hematologic CR (Complete Response)+ VGPR (very good partial response) at the completion of 6 cyels | 6 months
Rate of Hematologic ORR (Overall Response, CR+VGPR+low-dFLC response+PR) at the completion of 6 cyels | 6 months
Renal response at 6 months | 6 months
MRD status at 6 months | 6 months
Renal Survival in 2 years | 2 years
Overall Survival in 2 years | 2 years
TRAEs | 2 years
  Treatment-related adverse events up to 2 years

IPD SHARING:
Plan to Share IPD: No